CLINICAL TRIAL: NCT00894257
Title: Trends in Risk of Mother-to-child Transmission of Hepatitis C Through Analysis of Prevalence of Risk Factors for Maternal Infection Among a Southern European Population
Brief Title: Trends in Risk Factors for Mother-to-Child Transmission of Hepatitis C Among a Southern European Population
Acronym: EPIALHICE B
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Marine Barjoan Eugenia, CHU Nice
Other Study IDs: 07-PP-06
Record Dates: First submitted 2009-05-05; First posted 2009-05-06 (Estimated); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Hepatitis C Virus; HIV Infections; Pregnancy
Keywords: HCV infected pregnant women
MeSH Terms: conditions — Hepatitis C; HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HCV/HIV infected pregnant women

SUMMARY:
According to the centres taking part in the ALHICE survey, the number of HIV-HCV co-infected women is currently decreasing. This drop was first noted in 2006 and persisted in 2007. What might have been considered a chance phenomenon during the first year (2006) was confirmed in the beginning of 2008. In view of this information, the investigators wished to ascertain the reality of this trend and to investigate its causes, by attempting to answer the following questions: - Has the prevalence of risk factors for HCV infection changed among the general population over the past 10 years?

* Has the prevalence of risk factors for HCV infection changed among HIV/HCV co-infected women over the past 10 years?
* Is the change in the number of co-infected women who gave birth during the past 10 years related to the prevalence of certain risk factors among this population?
* Is the change in the number of co-infected women who gave birth during the past 10 years related to a decrease in certain risk factors for HCV infection among the general population?
* Have changes in addictive behaviour among women of child-bearing age played a role in the decreasing number of HCV-contaminated children? Furthermore, follow-up data from HCV-infected children born during this period will provide information concerning the course of HCV infection.

The objectives are to study trends in numbers of deliveries among HCV/HIV co-infected women as well as trends in risk factors for HCV infection among women of child bearing age and lastly to create a cohort of HCV infected children.

DETAILED DESCRIPTION:
Materials and Methods:

This multi-centre epidemiological study (CHU Nice, CHU Toulouse, CHU Montpellier, H Clinic Barcelona, H Mar Barcelona) consists in two parts. Our study does not interfere with the usual management of mother and child as laboratory data (virology, immunology, and liver function) are already included in the medical files. Data collection will be conducted via an anonymous questionnaire by an only one clinical research assistant who will travel to each participating centre. These data are contained in the mother's and child's medical files. The data concerning the socio-demographic characteristics of mother, the characteristics of HIV and HCV infection with special attention for infection risk factors, and the circumstances of the delivery. The questionnaire among children include laboratory results at birth, M6, and M12, as well as assessment of hepatic fibrosis.

Data were analysed using SPSS software. Qualitative variables were tested by Chi-square and Fisher's exact test. For quantitative variables, the non-parametric Mann-Whitney test was used (median, 25th and 75th quartile). A p-value inferior than 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Infected HIV/HCV pregnant women
* All women to give birth in 1 randomized week each 6 months

Ages: 15 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: HCV/HIV infected pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2009-05-25 (Actual); Primary Completion 2014-04-15 (Actual); Study Completion 2014-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugénia MARINE-BARJOAN, MD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (3):
- France (3):
  - CHU Montpellier, Montpellier
  - CHU Nice, Nice
  - CHU Toulouse, Toulouse